CLINICAL TRIAL: NCT04466683
Title: Phase II Protocol of Low-Dose Whole Thorax Megavoltage Radiotherapy for Patients With SARS-COV-2 Pneumonia
Brief Title: Low-Dose Radiotherapy For Patients With SARS-COV-2 (COVID-19) Pneumonia
Acronym: PREVENT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Arnab Chakravarti, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENT
Record Dates: First submitted 2020-06-20; First posted 2020-07-10 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Covid-19; Sars-CoV2; Pneumonia
Keywords: radiation; radiotherapy; Linac
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 to receive radiation therapy (2 different doses) or control (no radiation). Sixty subjects will be enrolled to 3 arms and the best dose chosen after enrolling 60 subjects. Randomization of an additional 40 subjects will be randomized 2:1 to receive radiation therapy (best dose) versus control with no radiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Low radiation arm (Experimental): A single dose of 35 cGY delivered to the whole thorax
  Interventions: Radiation: Low dose radiation 35 cGy
- High radiation arm (Experimental): A single dose of 100 cGY delivered to the whole thorax
  Interventions: Radiation: High dose radiation 100 cGy
- Control arm (No Intervention): Patients will receive no radiation therapy but will have research samples collected and best supportive care

INTERVENTIONS:
Radiation: Low dose radiation 35 cGy — A dose of 35 cGy of whole thorax irradiation will be delivered at a single timepoint
  Arms: Low radiation arm
Radiation: High dose radiation 100 cGy — A dose of 100 cGy of whole thorax irradiation will be delivered at a single timepoint
  Arms: High radiation arm

SUMMARY:
Low doses of radiation in the form of chest x-rays has been in the past to treat people with pneumonia. This treatment was thought to reduce inflammation and was found to be effective without side effects. However, it was an expensive treatment and was eventually replaced with less expensive treatment options like penicillin.

The COVID-19 virus has emerged recently, causing high rates of pneumonia in people. The authors believe that giving a small dose of radiation to the lungs may reduce inflammation and neutralize the pneumonia caused by COVID-19. For this study, the x-ray given is called radiation therapy. Radiation therapy uses high-energy X-ray beams from a large machine to target the lungs and reduce inflammation. Usually, it is given at much higher doses to treat cancers.

The purpose of this study is to find out if adding a single treatment of low-dose x-rays to the lungs might reduce the amount of inflammation in the lungs from COVID-19 infection, which could reduce the need for a ventilator or breathing tube.

DETAILED DESCRIPTION:
The authors propose a two-step randomized Phase II study to determine if single fraction low dose whole thorax megavoltage radiotherapy (LD-WTRT) can produce meaningful clinical benefit in COVID-19 patients. In Step 1, patients would be randomized 1:2 to standard of care without or with LD-WTRT. Patients randomized to LD-WTRT would be further randomized to either 35 cGy or 100 cGy. After 20 patients have been enrolled on each low-dose radiotherapy arm, they will be evaluated to determine the selection of the "best radiotherapy dose-arm" for the remainder of the patients. This will be done by analyzing clinical benefit, risk profile, and the dynamics of biomarker change, specifically focusing on IL-6

1. If the rate of Grade 4 toxicity is lower by an absolute rate of 15% when comparing the 35 cGy and 100 cGy arms, the arm with the lower toxicity rate will be used for Step 2 of the trial.
2. If the crude clinically meaningful event rate (CMER) which is a composite endpoint, is lower by an absolute rate of 20% when comparing the 35 cGy and 100 cGy arms, the lower CMER rate arm will be used for Step 2. CMER is defined as a composite of :

   1. Rate of mechanical ventilation (MV)
   2. Rate of prolonged hospital stay >10 days (PHS)
   3. Crude all-cause mortality rate at the time of analysis
3. If the crude CMER is < 20% difference between the 35 cGy and 100 cGy arms, the investigators will determine whether there is a trend suggesting less Facility Resource Utilization Rate (FRUR). If the FRUR is 20% lower in either the 35 cGy or 100 cGy arms, that dose will be used for Step 2. The FRUR is based upon:

   1. Days of mechanical ventilation
   2. Days of hospitalization.
4. If both crude CMER and FRU rates do not differ by at least 20%, the investigators will evaluate the area under the curve (AUC) for IL-6 levels drawn within 24 hours before LD-WTRT and at 48 hours (2d) and 168 hours (7d) after radiation. If one of the two arms has a 20% lower serum IL-6 AUC one week after radiotherapy, the investigators will select that arm for Step 2.
5. If none of the parameters in numbers 1-4 above differ in the criteria listed, the investigators will use the lower dose of 35 cGy for Step 2.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed diagnosis of SARS-CoV-2 pneumonia
* Currently hospitalized with COVID-19
* Symptomatic fever, cough and/or dyspnea for < 9 days
* Patient or legal/authorized representative can understand and sign the study informed consent document
* Able to be positioned on a linear-accelerator couch for Radiation Therapy delivery
* And at least one of the following risk factors for significant pulmonary compromise:

  1. Fever > 102 degrees Fahrenheit during index admission
  2. Respiratory rate of ≥ 26 / minute within 24 hours of screening
  3. SpO2 ≤ 95% on room air within 24 hours of screening
  4. Any patient requiring 4 L/min oxygen therapy to maintain SpO2 >93% within 24 hours of screening
  5. Ratio of partial pressure of arterial oxygen to fraction of inspired air < 320.
* Patients may be enrolled on this trial while concurrently enrolled on other COVID-19 clinical trials.

Exclusion Criteria:

* Currently requiring mechanical ventilation
* Prior thoracic radiotherapy, with the exception of the following:

  1. Breast or post-mastectomy chest wall radiation (without regional nodal irradiation) may be included at the discretion of the site primary investigator, and
  2. Thoracic skin radiation therapy (without regional nodal irradiation) is allowed.
* Known hereditary syndrome with increased sensitivity to radiotherapy, including ataxia-telangiectasia, xeroderma pigmentosum, and Nijmegen Breakage Syndrome
* Known prior systemic use of the following drugs: Bleomycin, Carmustine, Methotrexate, Busulfan, Cyclophosphamide, or Amiodarone
* History of or current diagnosis of pulmonary fibrosis, or an alternative pulmonary condition responsible for significant lung compromise at the discretion of the site primary investigator
* History of lung lobectomy or pneumonectomy
* Known history of pulmonary sarcoidosis, Wegener's granulomatosis, systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, polymyositis/dermatomyositis, Sjögren's syndrome, mixed connective tissue disease, Churg-Strauss syndrome, Goodpasture's syndrome, or ankylosing spondylitis.
* Symptomatic congestive heart failure within the past 6 months including during current hospitalization
* History of recent or current malignancy receiving any cytotoxic chemotherapy or immunotherapy within the past 6 months.
* History of bone marrow transplantation.
* History of any solid organ transplant (renal, cardiac, liver, lung) requiring immunosuppressive therapy.
* Females who are pregnant or breast feeding.
* Inability to undergo radiotherapy for any other medical or cognitive issues.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Step 1 Dose selection | At least 2 weeks after the 60th patient enrolled has been evaluated for adverse events. It is estimated that the time frame will be about 1 year to complete enrollment.
  The rate of grade 4 toxicity, the rate of mechanical ventilation, the rate of hospital stay greater than 10 days, and the crude all-cause mortality rate will be used to calculate the clinically meaningful event rate (CMER). The rates range would be from 0 to 100% with a lower rate indicating a more favorable dose.
Clinical benefit of Step 2 Radiation dose | up to 30 days from the last patient enrollment in Step 2 which is estimated to be about 2 years.
  Clinical benefit will have the composite endpoint with the following 3 elements: the rate of mechanical ventilation, the rate of hospital stays of greater than 10 days and the rate of all-cause mortality at 30 from enrollment. A lower rate would indicate a positive clinical benefit and would range from 0 to 100%

SECONDARY OUTCOMES:
Changes of the cost of care for the control arm versus the radiation arms | The discharge of the last patient enrolled is estimated to be about 2 years.
  Billing codes will be collected to determine the total cost of hospitalization for each patient at discharge. The cost of hospitalization for the control arm versus experimental radiation arms will be compared.

OTHER OUTCOMES:
Changes in lymphocyte count between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization.
  Compare differences within and between arms lymphocyte count in K/ul.
Changes in neutrophil count between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms neutrophil count in K/ul .
Changes in neutrophil to lymphocyte ratio between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms for the neutrophil to lymphocyte ratio. A decrease in the ratio of neutrophil to lymphocyte count would indicate a more favorable treatment outcome.
Changes in blood C-reactive protein between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms for the C-reactive protein in mg/L. A decrease in C-reactive protein value would indicate a more favorable treatment outcome.
Changes in blood IL-6 levels between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms for the IL-6 in pg/ml. A decrease in IL-6 value would indicate a more favorable treatment outcome.
Changes in blood D-Dimer levels between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms for the D-Dimer in mcg/ml. A decrease in D-Dimer value would indicate a more favorable treatment outcome.
Changes in blood Lactate dehydrogenase (LDH) levels between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms for the LDH in U/L. A decrease in LDH value would indicate a more favorable treatment outcome.
Changes in blood ferritin levels between control and experimental arms | Samples are collected pre-dose, 48-72 hours post radiation dose, and 7 days after radiation dose. Control subjects have blood samples collected post randomization, 48-72 hours post randomization, and 7 days post randomization
  Compare differences within and between arms for ferritin in ng/ml. A decrease in Ferritin value would indicate a more favorable treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Chakravarti, MD, Principal Investigator — James Cancer Hospital, Department of Radiation Oncology
Locations (7):
- United States (6):
  - Boca Raton Regional Hospital Lynn Cancer Institute, Boca Raton, Florida
  - Miami Cancer Institute, Miami, Florida
  - Loyola University Chicago, Maywood, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Lowell General Hospital Cancer Center, Lowell, Massachusetts
  - Ohio State University James Cancer Hospital, Columbus, Ohio
- Hospital Universitario San Ignacio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McClelland S 3rd, Miller AC, Williams MD, Anthony BP, Chakravarti A, Anthony PA. Low-dose whole thorax radiation therapy for COVID-19 pneumonia: inpatient onboarding process for a randomized controlled trial. Rep Pract Oncol Radiother. 2021 Dec 30;26(6):1057-1059. doi: 10.5603/RPOR.a2021.0112. eCollection 2021. PMID 34992881